CLINICAL TRIAL: NCT02266602
Title: Intra-Operative Radiotherapy After Breast Conserving Therapy in the Treatment of in Situ and Early Stage Breast Cancer
Brief Title: Intraoperative Radiation Therapy in Early Stage Breast Cancer
Acronym: IORTBreast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Principal Investigator, Michelle Yao, MD, Benaroya Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11143
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: IORT; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other): Patients treated with intraoperative radiation therapy at the time of partial mastectomy.
  Interventions: Radiation: Intraoperative Radiation Therapy

INTERVENTIONS:
Radiation: Intraoperative Radiation Therapy — Intraoperative radiation therapy at the time of partial mastectomy in early stage breast cancer
  Other Names: IORT

SUMMARY:
Single arm study to assess the effectiveness of single dose intraoperative radiation therapy in patient with in situ and early stage breast cancer.

DETAILED DESCRIPTION:
The purpose of this clinical study is to assess the effectiveness of IORT, using an electronic brachytherapy system, in patients with limited-volume in situ and early stage breast cancer, with endpoints of:

* Local recurrence in early stage breast cancer patients treated with IORT.
* Toxicity associated with IORT.
* Long-term disease-specific and overall survival
* Cosmetic results using the Harvard Scale at start and follow-up periods in patients treated with IORT.
* Quality of life in patients treated with IORT.
* Health care costs associated with IORT.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Age ≥ 45 years.
2. Clinical stage Tis, T1, T2 (≤ 3cm), N0, M0 (AJCC Classification).
3. Invasive ductal or lobular carcinoma, DCIS and/ or pleomorphic lobular carcinoma in situ.

Exclusion Criteria:

1. Scleroderma, systemic sclerosis and active lupus.
2. Participation in an investigational drug or device study.
3. Previous ipsilateral radiation to the thorax or breast.
4. Multifocal breast cancer.
5. Pregnant patients.
6. Patient not competent to provide informed consent.
7. Neoadjuvant systemic therapy.
8. Lymphovascular invasion on biopsy pathology

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-02; Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Local Disease Relapse | 10 years
  Patients are evaluated clinically at 3 months, 6 months, 9 months, 1 year and every six months for 10 years for disease recurrence. In addition to clinical exams, yearly mammograms and other imaging studies as deemed appropriate will be obtained to rule out recurrent disease. Recurrent disease will be defined as cancer recurrence within 2cm of site of original tumor bed (marked by surgical clips).

SECONDARY OUTCOMES:
Disease specific and overall survival | 10 years
  Disease specific and overall survival will be obtained for all patients in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janie Grumley, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States